CLINICAL TRIAL: NCT01782599
Title: Electronic Cigarettes and Reactivity to Smoking Cues
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mclean Hospital (Other)
Responsible Party: Principal Investigator, Scott Lukas, Professor of Psychiatry, HMS and Director, McLean Imaging Center, Mclean Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: E-cigarettes and Cues
Record Dates: First submitted 2013-01-30; First posted 2013-02-04 (Estimated); Last update posted 2024-01-05 (Actual); Status verified 2024-01

CONDITIONS: Nicotine Dependence
MeSH Terms: conditions — Tobacco Use Disorder | interventions — Electronic Nicotine Delivery Systems

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Dual nicotine patch and electronic cigarette (Experimental): Nicotine patch and the electronic cigarette will be administered.
  Interventions: Other: Dual nicotine patch and electronic cigarette

INTERVENTIONS:
Other: Dual nicotine patch and electronic cigarette

SUMMARY:
The purpose of this study is to determine whether electronic cigarettes can reduce reactivity to smoking-related cues.

DETAILED DESCRIPTION:
Tobacco-related illness causes over 5 million deaths per year in the developed world, and most currently available smoking cessation treatments do not effectively enhance long-term cessation outcomes. Reactivity to smoking cues is one factor associated with relapse vulnerability, which is untreated by cessation aids such as NRT. Combining treatments, which ameliorate both pharmacological nicotine withdrawal and reduce smoking cue reactivity, may enhance smoking cessation success. During this study we will test whether combining NRT with non-nicotine containing electronic cigarettes (e-cigarettes) effectively reduces reactivity to smoking cues. The only source of nicotine participants will receive during the study will come from NRT. We will use e-cigarettes that provide no nicotine, yet may provide a similar experience to smoking as e-cigarettes taste and feel similar to a regular cigarette. However, since nicotine delivery is not associated with the act of smoking the reinforcing effects associated with smoking behavior may be reduced. Reactivity to smoking cues will be assessed using a battery of measures including: self-report, behavioral, and neuroimaging.

ELIGIBILITY:
Inclusion Criteria:

1. Provide written informed consent.
2. Be aged 18-45.
3. Report smoking cigarettes daily in the past 6 months.
4. Have expired breath CO indicative of regular smoking.
5. Have a score greater than 0 on the FTND.
6. Be willing to use Nicotine Replacement Therapy (NRT) and the e-cigarette for a period of 2 to 3 weeks.
7. Speak and read English.
8. Pass an MRI safety screen and meet inclusion criteria for MRI scans.

Exclusion Criteria:

1. Be pregnant (measured via urinalysis).
2. Meet current abuse or dependence criteria for any substance other than nicotine or caffeine (measured via the SCID 5).
3. Produce a positive urine screen for drugs of abuse or alcohol at the fMRI scan visits.
4. Meet DSM-IV criteria for major depressive episode in the past six months, lifetime DSM-IV diagnosis of organic mental disorder, schizophrenia, schizoaffective disorder, bipolar disorder, delusional disorder or psychotic disorders not elsewhere classified (measured via the SCID 5).
5. Be currently suicidal as assessed by DSM 5 and the Beck Depression Inventory.
6. Current use of medications or any history of a medical condition that might affect the central nervous system at the time of scanning including: Abnormal structural MRI, or a history of head trauma or injury causing loss of consciousness lasting longer than 3 minutes or associated with skull fracture or intracranial bleeding or who had irremovable magnetically active objects on or within their body, history of epilepsy, current use of a beta-blocker or prescription analgesic/anxiolytic. (assessed by self-report).
7. MRI exclusion criteria. (additional information outlined in the "protection of human subjects" section).
8. History of claustrophobia.
9. History of propylene glycol sensitivity/allergy.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 125 (Estimated)
Dates: Start 2013-01; Primary Completion 2024-10-01 (Estimated); Study Completion 2024-10-01 (Estimated)

PRIMARY OUTCOMES:
Reduction in Cue Reactivity | 2 weeks after use
  Outcomes will be measured using a battery of self-report, neuroimagning, and behavioral measures of cue-reactivity.

CONTACTS AND LOCATIONS:
Overall Officials: Amy C Janes, PhD, Principal Investigator — Mclean Hospital
Locations (1):
- Mclean Hospital Imaging Center, Belmont, Massachusetts, United States

REFERENCES:
- [Background] Janes AC, Pizzagalli DA, Richardt S, deB Frederick B, Chuzi S, Pachas G, Culhane MA, Holmes AJ, Fava M, Evins AE, Kaufman MJ. Brain reactivity to smoking cues prior to smoking cessation predicts ability to maintain tobacco abstinence. Biol Psychiatry. 2010 Apr 15;67(8):722-9. doi: 10.1016/j.biopsych.2009.12.034. Epub 2010 Feb 20. PMID 20172508
- [Background] Janes AC, Frederick Bd, Richardt S, Burbridge C, Merlo-Pich E, Renshaw PF, Evins AE, Fava M, Kaufman MJ. Brain fMRI reactivity to smoking-related images before and during extended smoking abstinence. Exp Clin Psychopharmacol. 2009 Dec;17(6):365-73. doi: 10.1037/a0017797. PMID 19968401